CLINICAL TRIAL: NCT03815097
Title: Prospective Study to Evaluate Mapleson Circuit With Monitored Anesthesia Care During EBUS Bronchoscopy
Brief Title: Prospective Study to Evaluate Mapleson Circuit With Monitored Anesthesia Care During Endobronchial Ultrasound (EBUS) Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CooperHS
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Adenopathy; Localized; Lung Cancer
MeSH Terms: conditions — Lymphadenopathy; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized study. The study will not be blinded. Subjects will be recruited from those who are referred to the interventional pulmonary department for EBUS bronchoscopy and who will be undergoing monitored anesthesia care (MAC) for their procedure. Subjects will then be randomized (via an computer randomizing algorithm) to receive conventional MAC vs. MAC with a mapleson circuit and nasal trumpet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Monitored anesthesia care with a mapleson circuit and nasal trumpet
  Interventions: Procedure: Mapleson circuit and nasal trumpet
- Standard of care (No Intervention): Standard monitored anesthesia care

INTERVENTIONS:
Procedure: Mapleson circuit and nasal trumpet — The Mapleson Circuit is a breathing system used to deliver oxygen and remove carbon dioxide during anesthesia. It consists of fresh oxygen flow, a reservoir bag, an expiratory valve, tubing, and a connection to the patient. There are different types of Mapleson circuits depending on the different arrangements of its components. We plan to use a Mapleson D circuit attached to a nasal trumpet via a connector.
  Arms: Intervention

SUMMARY:
If the investigators can prove that the use of a mapleson circuit attached to a nasal trumpet employed during monitored anesthesia care leads to less sedation requirements, less procedure interruptions, shorter procedure duration, this would allow for to standardization of the type of anesthetic employed for EBUS at the investigators' institution and elsewhere. Less hypoxic episodes and less anesthetic requirements would benefit outcomes, lead to less recovery time and earlier discharges. Shorter procedural duration will create greater efficiency in the short procedure unit where the EBUS are performed.

DETAILED DESCRIPTION:
Monitored anesthesia Care (MAC) is a type of conscious sedation delivered by an anesthesiologist, during which different medications are given, usually via the intravenous route, to obtain varying levels of sedation depending on the surgery or procedure. This is routinely done for all EBUS procedures at Cooper University Hospital. Since MAC anesthesia does not include having a secure airway, occasionally the patient may develop episodes in which their oxygen level drops. During these episodes, the anesthesiologist will stop the procedure temporarily until the oxygen level returns to a normal range.

Often, changes in sedation amount is also required during this time. In traditional MAC anesthesia, the patient is receiving oxygen via a nasal cannula or a mask capable of measuring capnography. If oxygen is delivered via a capnography mask, the routine is to create a hole with scissors in the side of the mask in order to allow the bronchoscope into the patient's mouth. The Mapleson Circuit is a breathing system used to deliver oxygen and remove carbon dioxide during anesthesia. It consists of fresh oxygen flow, a reservoir bag, an expiratory valve, tubing, and a connection to the patient. There are different types of Mapleson circuits depending on the different arrangements of its components. The investigators plan to use a Mapleson D circuit attached to a nasal trumpet via a connector.

Endobronchial Ultrasound is a technique that uses ultrasound along with bronchoscopy to visualize the airway wall and structures adjacent to it. The clinical application and diagnostic benefits of EBUS have been well established, including diagnosis and staging of lung cancer. EBUS is usually performed under conscious sedation for patient comfort.

The route of entry for the EBUS scope requires passage through the vocal cords and into the airways. The procedure tends to be very stimulating for this reason, which is the reason for the necessity for anesthesia. Due to the amount of anesthesia required to subdue the airway reflexes for a smooth procedure, occasionally, the patient may become apneic or obstruct and not take adequate tidal volume breaths, leading to hypoxia. During these instances, the procedure is halted until the patient's oxygen levels return to baseline. The investigators have noticed that anesthesiologists who prefer to use the mapleson circuit with a nasal trumpet in place tend to less often interrupt the procedure due to hypoxia.

Placing a nasal trumpet in one nare allows access to the oropharynx, bypassing soft tissue that may relax under anesthesia and cause obstruction. Connecting that nasal trumpet to a device that can not only deliver oxygen efficiently when the subject is spontaneously breathing, but can also be used as an assist device to deliver assisted breaths in the event that the patient becomes hypoxic or apneic provides a method to oxygenate into the oropharynx without having to interrupt the procedure. It also helps maintain an airway from the nares into the oropharynx and prevent episodes of obstruction, which are commonly seen under MAC anesthesia. All anesthesiologists are familiar with the mapleson circuits as well as nasal trumpets.

No research has been done in this field specifically regarding EBUS. There is no anesthetic standard of care that is specific for an EBUS procedure. The anesthesia can be local anesthesia alone, with just topicalization of the airways, or MAC, or even general anesthesia with an endotracheal tube or a laryngeal mask airway. The choice is practitioner dependent.

Our experience has been that MAC with a mapleson circuit leads to less procedural interruptions, less hypoxic episodes and shorter procedural duration.

ELIGIBILITY:
Inclusion Criteria:

1. Age> 18
2. Patient undergoing EBUS bronchoscopy
3. Patient undergoing moderate conscious sedation

Exclusion Criteria:

1. Subjects age <18
2. Subjects requiring general anesthesia
3. Subjects with previous nasal surgeries
4. Subjects with Oxygen saturation < 90% on room air prior to procedure
5. Subjects who are pregnant
6. Subjects with known facial fractures or recent facial trauma
7. Subjects on any anticoagulation that cannot be discontinued prior to the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2015-10-30 (Actual); Study Completion 2015-10-30 (Actual)

PRIMARY OUTCOMES:
Number of Interruptions of the procedures for any respiratory events | 2 years
  An interruption is defined as any respiratory event that requires an intervention by the anesthesia provider or one requiring the procedural physician to temporarily stop the procedure.

IPD SHARING:
Plan to Share IPD: No